CLINICAL TRIAL: NCT00871260
Title: Stress Testing and Cardiac Magnetic Resonance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16570B
Record Dates: First submitted 2009-03-24; First posted 2009-03-30 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; Stress Testing; Lexiscan (regadenoson); Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Coronary Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Other): Approximately 25 healthy volunteers will be recruited as controls. Scan will be done with regadenoson contrast.
  Interventions: Drug: regadenoson

INTERVENTIONS:
Drug: regadenoson — Subjects in open label group will be given a single dose of regadenoson (0.4 mg, i.e. 5 ml i.v. bolus) as contrast.
  Other Names: Lexiscan

SUMMARY:
The purpose of this study is to better define the role of a comprehensive stress MRI (which includes myocardial perfusion imaging, optimized coronary imaging, and myocardial scar imaging) in medical practice and in patient health management. Information gathered from the healthy volunteers that participate in this study will be compared to information from the coronary artery disease patients in this study in order to help further our understanding.

DETAILED DESCRIPTION:
Coronary artery disease is a major cause of morbidity and mortality in the United States. Currently, the presence of physiologically significant coronary disease is most commonly diagnosed using non-invasive imaging tests such as a nuclear stress test or an echo stress test. Unfortunately, nuclear stress tests require the use of ionizing radiation and have a limited spatial resolution. On the other hand, echo stress tests are dependent of adequate imaging windows. Adenosine stress testing combined with cardiac magnetic resonance (CMR) is a rapidly evolving technique for diagnosing significant coronary disease. It does not use ionizing radiation and has excellent image quality. In a recent meta-analysis of 14 studies with a total of 1,183 patients, the sensitivity and specificity of stress CMR for detecting significant coronary disease was 91% and 81%. Additionally, 2 studies have shown that patients with a normal stress CMR study have a <1% risk of having a cardiovascular event during the ensuing year. Another important advantage to stress CMR is the ability to fully quantify myocardial blood flow which may improve the diagnostic accuracy of stress CMR. In addition to perfusion imaging, CMR can directly visualize the coronary arteries, detect extremely small myocardial infarctions, and precisely measure the left ventricular function.

Although adenosine stress CMR is a rapidly maturing test, several important challenges exist. First, many patients find it difficult to tolerate the common side effects of adenosine in the confined space of the MRI scanner. Secondly, many patients under the influence of adenosine and its side effects cannot adequately hold their breath during image acquisition making image interpretation more difficult and quantitative analysis very time consuming. Finally, because adenosine must be continuously infused during a contrast-enhanced stress CMR, 2 separate intravenous (I.V.) catheters are needed. Most of the undesirable effects of adenosine are mediated through the adenosine A(2B) and A(3) receptors; where as, its desired vasodilator effects are mediated through the A(2A) receptor. The FDA recently approved an adenosine A(2A) receptor specific stress testing agent called regadenoson which is administered as a 10 second bolus and has an improved side effect and safety profile when compared to adenosine. With its improved tolerability and ease of use, regadenoson is a more ideal stress testing agent to use with CMR.

The purpose of this study is to determine whether a comprehensive regadenoson stress cardiac magnetic resonance study which includes myocardial perfusion imaging, optimized coronary imaging, and myocardial scar imaging provides incremental prognostic information over a clinical evaluation that includes nuclear stress testing.

ELIGIBILITY:
Inclusion Criteria:

* Suspected coronary artery disease
* Symptoms of possible coronary artery disease

Exclusion Criteria:

* Acute ST-elevation myocardial infarction
* Second or third degree AV block
* Severe Renal Disease (Glomerular Filtration Rate (GFR) <30cc/min or hemodialysis)
* Contra-indications to MRI (i.e. Implantable Cardioverter Defibrillator (ICD), pacemaker, aneurysm clip, etc)
* Hemodynamic instability
* Inability to provide informed consent
* Severe claustrophobia
* Pregnancy
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06-04 (Actual); Study Completion 2014-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Patel, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hachamovitch R, Berman DS, Shaw LJ, Kiat H, Cohen I, Cabico JA, Friedman J, Diamond GA. Incremental prognostic value of myocardial perfusion single photon emission computed tomography for the prediction of cardiac death: differential stratification for risk of cardiac death and myocardial infarction. Circulation. 1998 Feb 17;97(6):535-43. doi: 10.1161/01.cir.97.6.535. PMID 9494023
- [Background] McCrohon JA, Lyne JC, Rahman SL, Lorenz CH, Underwood SR, Pennell DJ. Adjunctive role of cardiovascular magnetic resonance in the assessment of patients with inferior attenuation on myocardial perfusion SPECT. J Cardiovasc Magn Reson. 2005;7(2):377-82. doi: 10.1081/jcmr-200053627. PMID 15881517
- [Background] Nandalur KR, Dwamena BA, Choudhri AF, Nandalur MR, Carlos RC. Diagnostic performance of stress cardiac magnetic resonance imaging in the detection of coronary artery disease: a meta-analysis. J Am Coll Cardiol. 2007 Oct 2;50(14):1343-53. doi: 10.1016/j.jacc.2007.06.030. Epub 2007 Sep 17. PMID 17903634
- [Background] Jahnke C, Nagel E, Gebker R, Kokocinski T, Kelle S, Manka R, Fleck E, Paetsch I. Prognostic value of cardiac magnetic resonance stress tests: adenosine stress perfusion and dobutamine stress wall motion imaging. Circulation. 2007 Apr 3;115(13):1769-76. doi: 10.1161/CIRCULATIONAHA.106.652016. Epub 2007 Mar 12. PMID 17353441
- [Background] Ingkanisorn WP, Kwong RY, Bohme NS, Geller NL, Rhoads KL, Dyke CK, Paterson DI, Syed MA, Aletras AH, Arai AE. Prognosis of negative adenosine stress magnetic resonance in patients presenting to an emergency department with chest pain. J Am Coll Cardiol. 2006 Apr 4;47(7):1427-32. doi: 10.1016/j.jacc.2005.11.059. Epub 2006 Mar 20. PMID 16580532
- [Background] Schwitter J, Wacker CM, van Rossum AC, Lombardi M, Al-Saadi N, Ahlstrom H, Dill T, Larsson HB, Flamm SD, Marquardt M, Johansson L. MR-IMPACT: comparison of perfusion-cardiac magnetic resonance with single-photon emission computed tomography for the detection of coronary artery disease in a multicentre, multivendor, randomized trial. Eur Heart J. 2008 Feb;29(4):480-9. doi: 10.1093/eurheartj/ehm617. Epub 2008 Jan 21. PMID 18208849
- [Background] Hachamovitch R, Hayes SW, Friedman JD, Cohen I, Berman DS. Comparison of the short-term survival benefit associated with revascularization compared with medical therapy in patients with no prior coronary artery disease undergoing stress myocardial perfusion single photon emission computed tomography. Circulation. 2003 Jun 17;107(23):2900-7. doi: 10.1161/01.CIR.0000072790.23090.41. Epub 2003 May 27. PMID 12771008
- [Background] Wang L, Jerosch-Herold M, Jacobs DR Jr, Shahar E, Detrano R, Folsom AR; MESA Study Investigators. Coronary artery calcification and myocardial perfusion in asymptomatic adults: the MESA (Multi-Ethnic Study of Atherosclerosis). J Am Coll Cardiol. 2006 Sep 5;48(5):1018-26. doi: 10.1016/j.jacc.2006.04.089. Epub 2006 Aug 17. PMID 16949496
- [Background] Patel AR, Epstein FH, Kramer CM. Evaluation of the microcirculation: advances in cardiac magnetic resonance perfusion imaging. J Nucl Cardiol. 2008 Sep-Oct;15(5):698-708. doi: 10.1016/j.nuclcard.2008.07.002. No abstract available. PMID 18761273
- [Background] Sakuma H, Ichikawa Y, Chino S, Hirano T, Makino K, Takeda K. Detection of coronary artery stenosis with whole-heart coronary magnetic resonance angiography. J Am Coll Cardiol. 2006 Nov 21;48(10):1946-50. doi: 10.1016/j.jacc.2006.07.055. Epub 2006 Oct 31. PMID 17112982
- [Background] Wagner A, Mahrholdt H, Holly TA, Elliott MD, Regenfus M, Parker M, Klocke FJ, Bonow RO, Kim RJ, Judd RM. Contrast-enhanced MRI and routine single photon emission computed tomography (SPECT) perfusion imaging for detection of subendocardial myocardial infarcts: an imaging study. Lancet. 2003 Feb 1;361(9355):374-9. doi: 10.1016/S0140-6736(03)12389-6. PMID 12573373
- [Background] Bellenger NG, Davies LC, Francis JM, Coats AJ, Pennell DJ. Reduction in sample size for studies of remodeling in heart failure by the use of cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2000;2(4):271-8. doi: 10.3109/10976640009148691. PMID 11545126
- [Background] Lieu HD, Shryock JC, von Mering GO, Gordi T, Blackburn B, Olmsted AW, Belardinelli L, Kerensky RA. Regadenoson, a selective A2A adenosine receptor agonist, causes dose-dependent increases in coronary blood flow velocity in humans. J Nucl Cardiol. 2007 Jul;14(4):514-20. doi: 10.1016/j.nuclcard.2007.02.016. PMID 17679059
- [Background] Ding S, Wolff SD, Epstein FH. Improved coverage in dynamic contrast-enhanced cardiac MRI using interleaved gradient-echo EPI. Magn Reson Med. 1998 Apr;39(4):514-9. doi: 10.1002/mrm.1910390403. PMID 9543412
- [Background] Christian TF, Rettmann DW, Aletras AH, Liao SL, Taylor JL, Balaban RS, Arai AE. Absolute myocardial perfusion in canines measured by using dual-bolus first-pass MR imaging. Radiology. 2004 Sep;232(3):677-84. doi: 10.1148/radiol.2323030573. Epub 2004 Jul 29. PMID 15284436
- [Background] Mor-Avi V, Akselrod S, David D, Keselbrener L, Bitton Y. Myocardial transit time of the echocardiographic contrast media. Ultrasound Med Biol. 1993;19(8):635-48. doi: 10.1016/0301-5629(93)90070-5. PMID 8134968
- [Background] Jerosch-Herold M, Wilke N, Stillman AE. Magnetic resonance quantification of the myocardial perfusion reserve with a Fermi function model for constrained deconvolution. Med Phys. 1998 Jan;25(1):73-84. doi: 10.1118/1.598163. PMID 9472829
- [Background] Spuentrup E, Katoh M, Buecker A, Manning WJ, Schaeffter T, Nguyen TH, Kuhl HP, Stuber M, Botnar RM, Gunther RW. Free-breathing 3D steady-state free precession coronary MR angiography with radial k-space sampling: comparison with cartesian k-space sampling and cartesian gradient-echo coronary MR angiography--pilot study. Radiology. 2004 May;231(2):581-6. doi: 10.1148/radiol.2312030451. Epub 2004 Mar 24. PMID 15044745
- [Background] Diamond GA, Forrester JS. Analysis of probability as an aid in the clinical diagnosis of coronary-artery disease. N Engl J Med. 1979 Jun 14;300(24):1350-8. doi: 10.1056/NEJM197906143002402. PMID 440357
- [Background] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226
- [Derived] Bhave NM, Freed BH, Yodwut C, Kolanczyk D, Dill K, Lang RM, Mor-Avi V, Patel AR. Considerations when measuring myocardial perfusion reserve by cardiovascular magnetic resonance using regadenoson. J Cardiovasc Magn Reson. 2012 Dec 28;14(1):89. doi: 10.1186/1532-429X-14-89. PMID 23272658

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Patients: Twenty healthy subjects underwent CMR perfusion imaging during resting conditions, during regadenoson-induced hyperemia (0.4 mg), and after 15 min of recovery.
Period: Overall Study
Arm/Group | Healthy Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty healthy subjects underwent CMR perfusion imaging during resting conditions, during regadenoson-induced hyperemia (0.4 mg), and after 15 min of recovery.
Groups:
- Healthy Patients: Due to low enrollment, twenty healthy subjects underwent CMR perfusion imaging during resting conditions, during regadenoson-induced hyperemia (0.4 mg), and after 15 min of recovery. All analyzes were based upon current enrollment.
Arm/Group | Healthy Patients
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12
  Not Caucasian | 8

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiovascular Events
Description: Major adverse cardiovascular events, such as death, myocardial infarction, unstable angina, congestive heart failure, or cerebral vascular accident.
Time Frame: 3 years
Population: All efforts were taken to gather all possible data but none were obtained for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 20
Participants | 0

2. Secondary Outcome: Relationship Between SPECT and CMR Results of Myocardial Perfusion Imaging
Description: Relationship between SPECT and CMR results of myocardial perfusion imaging for 1 Year
Time Frame: 1 year
Population: Coronary imaging pulse sequences were unable to be performed. All efforts were taken to gather all possible data but none were obtained for this Outcome Measure.
Arm/Group | Healthy Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Optimization of Coronary Imaging Using CMR
Description: Optimization of coronary imaging using CMR for 1 Year
Time Frame: 1 year
Population: Coronary imaging were unable to be performed. All efforts were taken to gather all possible data but none were obtained for this Outcome Measure.
Arm/Group | Healthy Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 Years
Description: Patients were assessed at clinic for medication compliance and self-reported medication side effects, in addition to follow-up calls for any additional medication side effects.
Arm/Group | Healthy Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Patients (N=20)
Dyspnea or difficulty with breath (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Palpitations (Cardiac disorders) | 7 (7)
Chest pressure or heaviness (Cardiac disorders) | 7 (7)
Flushing (Cardiac disorders) | 5 (5)
Dysgeusia immediately following aminophylline administration (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was conducted in a small number of healthy volunteers. We could not assess whether a rest stress protocol as opposed to a stress-recovery protocol would mask the presence of ischemia due to contrast contamination of stress images. It is possible that postregadenoson recovery imaging either earlier or later would have demonstrated a lesser degree of residual hyperemia. It is unknown whether a relatively modest underestimation of perfusion reserve would have clinical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No